CLINICAL TRIAL: NCT02975973
Title: Prefrontal Cortical Engagement Through Non-Invasive Brain Stimulation in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Raymond Cho, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-41815
Record Dates: First submitted 2016-11-23; First posted 2016-11-29 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Schizophrenia; Psychosis
Keywords: tDCS; cognitive control; EEG; gamma oscillations
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- 2.5mA (Experimental): Active stimulation group will receive 20 minutes of 2.5 mA transcranial direct current stimulation.
  Interventions: Device: transcranial direct current stimulation
- 2.0mA (Experimental): Active stimulation group will receive 20 minutes of 2.0 mA transcranial direct current stimulation.
  Interventions: Device: transcranial direct current stimulation
- 1.5mA (Experimental): Active stimulation group will receive 20 minutes of 1.5 mA transcranial direct current stimulation.
  Interventions: Device: transcranial direct current stimulation
- 0mA (Sham Comparator): This will be an active sham involving transcranial direct current stimulation, though stimulation will be brief (15 msec) and have low current (0.11 mA) pulses every 550 ms.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — transcranial direct current stimulation (tDCS) is a safe, noninvasive, weak electrical current delivery that stimulates brain function. It is a novel therapeutic for cognition in schizophrenia.

SUMMARY:
Cognitive impairments in schizophrenia are the most debilitating aspect of the illness and poorly treated by current medications. This study investigates transcranial direct current stimulation (tDCS) - a safe, noninvasive weak electrical current delivery to stimulate brain function - as a novel therapeutic for cognition in schizophrenia. Integrating neurostimulation, electrophysiology and neuroimaging, this project aims to study tDCS effects on cognition by verifying therapeutic target engagement, evaluating the tolerability of tDCS sessions, and optimizing treatment parameters.

DETAILED DESCRIPTION:
Cognitive deficits are a strong predictor of functional outcome in schizophrenia, yet poorly remediated by current treatments. Disturbances in dorsolateral prefrontal cortex (DLPFC) function underlie core impairments such as in cognitive control and thus represent a critical target for novel therapeutics. Initial studies indicate transcranial direct-current stimulation (tDCS) may be effective in reducing symptoms due to DLPFC dysfunction. While tDCS potentially represents an exciting, novel therapeutic advance, a number of basic questions should be addressed prior to conducting larger-scale clinical trials, including: verifying therapeutic target engagement, optimizing treatment parameters, and evaluating for meaningful clinical effects. Recent studies employing tDCS to enhance prefrontal cortical function in schizophrenia applied stimulating electrodes over the left frontal scalp region, putatively targeting the left DLPFC. However, explicit confirmation of such target engagement is lacking. Further, EEG studies have demonstrated close links of frontal cortical gamma oscillations to cognitive control processes but modulation of this critical physiologic process has not been investigated. Accordingly, the primary aim of this study is to employ multimodal imaging to explicitly test for the assumed DLPFC engagement (fMRI) and modulation of frontal gamma activity (EEG) by tDCS. This study will also investigate the optimization of tDCS application parameters. Analogous to dose-finding investigations in drug studies, we will conduct a parametric investigation of optimal current strengths. Also, while there is extensive evidence for tolerability of single session tDCS, confirmation of feasibility of multisession optimized protocols in schizophrenia is lacking and so will be explicitly evaluated.

In summary, a successful outcome of this study would provide tDCS the sound mechanistic and methodologic basis for more definitive testing in large-scale clinical trials as a highly innovative therapeutic intervention for cognitive impairments in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-35 years;
2. within first five years of antipsychotic treatment;
3. on stable doses of antipsychotic medication for at least one month;
4. Clinically stable as defined by Clinical Global Impression-Severity scale (CGI-S) less than or equal to 4 (moderately ill);
5. Mild to severe cognitive impairment in MATRICS Consensus Cognitive Battery (composite scores <40);
6. DSM-5 MINI 7.0.2 criteria for schizophrenia or schizoaffective by patient SCID

Exclusion Criteria:

1. Mental retardation as defined by pre-morbid IQ by Wechsler Test of Adult Reading at screening <70 or Spanish Word Accentuation Test;
2. significant head injury;
3. History of severe medical or neurological illnesses
4. pregnancy or postpartum (<6 weeks after delivery or miscarriage);
5. inability to provide informed consent;
6. significant color blindness that affects task performance;
7. Positive urine drug screen (exception for marijuana) or presence of substance use disorder within 1 month;
8. Currently on benzodiazepines or mood stabilizers affecting GABA

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-11; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Cho, M.D., M.Sc., Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be open to sharing after primary findings of study have been published

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The reason we have fewer subjects randomized than enrolled is that some participants did not meet criteria to be randomized. These subjects were consented and completed many assessments, but were ultimately not randomized due to how they scored on some assessments. For instance, some peoples MCCB score was too high to be randomized into the study.
Pre-assignment Details: The primary reasons for ineligibility were not meeting the early psychosis criterion (< 5 years of treatment), not taking any medication, and drug use. There were also many who did not even enter screening due to the assessment that they would highly likely not meet the threshold of requirement cognitive impairment (MATRICS score 40).
Groups:
- 0mA (Active Placebo): This will be an active sham involving transcranial direct current stimulation, though stimulation will be brief (15 msec) and have low current (0.11 mA) pulses every 550 ms.
  transcranial direct current stimulation: transcranial direct current stimulation (tDCS) is a safe, noninvasive, weak electrical current delivery that stimulates brain function. It is a novel therapeutic for cognition in schizophrenia.
Period: Overall Study
Arm/Group | 2.5mA | 2.0mA | 1.5mA | 0mA (Active Placebo)
Started | 1 | 2 | 1 | 4
Completed | 0 | 1 | 0 | 4
Not Completed | 1 | 1 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5mA | 2.0mA | 1.5mA | 0mA (Active Placebo) | Total
Number analyzed (Participants) | 1 | 2 | 1 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 1 | 4 | 8
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22 (0) | 26 (3.65) | 22 (0) | 23 (2.44) | 24 (2.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 2
  Male | 1 | 2 | 0 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 3 | 5
  White | 0 | 1 | 0 | 1 | 2
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 1 | 4 | 8
MCCB Score [Mean (Standard Deviation); unit: units on a scale] — Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB).
  Intended to provide a relatively brief evaluation of key cognitive domains that are relevant to schizophrenia and related disorders, the battery is appropriate for use as an outcome measure for clinical trials of cognition-enhancing drugs, when studying cognitive remediation, to measure cognitive change, and as a cognitive reference point for nonintervention studies of schizophrenia and other severe psychiatric disorders.
  Higher scores are better.
  units on a scale | 15 (0) | 17.5 (4.95) | 35 (0) | 32 (12.72) | 26.6 (11.94)

OUTCOME MEASURES:

1. Primary Outcome: tDCS Engagement of DLPFC Activity Indexed by fMRI BOLD Imaging
Description: Change from Baseline to week 1 as measured by modulation of fMRI BOLD signal in DLPFC in the context of cognitive control task performance.
Time Frame: 1 week
Population: Our analytic strategy involved defining regions of interest (ROI) derived from group averages across all study subjects but due to unforeseen circumstances, we recruited far too few subjects to derive meaningful group averages. Individual subject and by extension, condition-specific averages that are based on such ROIs, could therefore not be derived. However, we will upload our raw data to the National Data Archive to be accessed for any potential analyses with data pooled from other studies.
Arm/Group | 2.5mA | 2.0mA | 1.5mA | 0mA (Active Placebo)
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: tDCS Engagement of DLPFC Activity Indexed by Modulation of Frontal Cortical Gamma Oscillations
Description: Change from Baseline to week 1 as measured by EEG frontal gamma oscillations in the context of cognitive control task performance
Time Frame: 1 week
Population: as for outcome 1
Arm/Group | 2.5mA | 2.0mA | 1.5mA | 0mA (Active Placebo)
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Optimal tDCS Strength for DLPFC Engagement
Description: Change from baseline to 1 week in DLPFC engagement across conditions (1.5 vs 2.0 vs 2.5 mA)
Time Frame: 1 Week
Population: as for outcome 1
Arm/Group | 2.5mA | 2.0mA | 1.5mA | 0mA (Active Placebo)
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Tolerability and Feasibility of Multi-session tDCS in Schizophrenia
Description: The percentage of participants able to complete the full study.
Time Frame: 1 week
Population: Due to unforeseen circumstances, we were unable to sufficiently recruit enough subjects to complete the originals plans for analysis. The percentages below are the percent of subjects who completed each condition.
Measure: Number; unit: percentage of participants completed
Arm/Group | 2.5mA | 2.0mA | 1.5mA | 0mA (Active Placebo)
Number analyzed (Participants) | 1 | 2 | 1 | 4
percentage of participants completed | 0 | 50 | 0 | 100

ADVERSE EVENTS:
Time Frame: Two Weeks
Arm/Group | 2.5mA | 2.0mA | 1.5mA | 0mA (Active Placebo)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2 | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 0/1 | 1/2 | 0/1 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5mA (N=1) | 2.0mA (N=2) | 1.5mA (N=1) | 0mA (Active Placebo) (N=4)
Exacerbation of Psychotic Symptoms (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5mA (N=1) | 2.0mA (N=2) | 1.5mA (N=1) | 0mA (Active Placebo) (N=4)
Minor Burn (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Minor burn at location of tDCS electrode placement.

LIMITATIONS AND CAVEATS:
Despite concerted and exhaustive subject recruitment efforts, the total number of patients completing the protocol was minimal. As such the sample size was inadequate for deriving any meaningful descriptive statistics or statistical comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT02975973/Prot_SAP_000.pdf